CLINICAL TRIAL: NCT06517446
Title: Effect of Optokinetic Virtual Reality Stimulation in Unilateral Vestibular Hypofunction Patients
Brief Title: Optokinetic Virtual Reality Stimulation in Unilateral Vestibular Hypofunction
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Ebru Sever, Specialist Physiotherapist, Medipol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EBRUDOKTORA
Record Dates: First submitted 2024-07-08; First posted 2024-07-24 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Vestibular Hypofunction
Keywords: Unilateral Vestibular Hypofunction; Virtual Reality; Optokinetic stimulation; Motion Sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (VR Group) (Experimental): Participants will receive a structured conventional vestibular rehabilitation program for eight weeks, once a week, in 45-minute sessions supervised by a physiotherapist. The program will be individualized based on Cawthorne-Cooksey exercises and progressively advanced with the guidance of a vestibular therapist. Additionally, participants will be provided with a home exercise program, to be performed twice daily (morning and evening), with 10 repetitions each time.
  Interventions: Other: Conventional rehabilitation program based on Cawthorne Cooksey exercises
- Group 2 (OKS Group) (Experimental): Optokinetic stimulation sessions are planned with a balloon rotation speed of 20°/s (degrees per second) during the first four weeks. In the fifth and sixth weeks, the speed will be increased to 25°/s, and in the seventh and eighth weeks, it will be raised to 30°/s. The background screen will be set to rotate in the same direction as the balloons, with a rotation speed equal to 30-50% of the balloon rotation speed. The visual stimulus scene will feature colorful balloons moving in circular patterns, both clockwise and counterclockwise. Participants will be instructed to focus on a red balloon within the scene. The initial session duration will be set at 30 seconds and will be gradually increased up to 150 seconds depending on the participant's tolerance. Each session will include three repetitions of optokinetic stimulation.
  Interventions: Other: Optokinetic Virtual Reality Stimulation
- Group 3 (VR+OKS Group) (Experimental): Participants in this group will receive both the vestibular rehabilitation program and the optokinetic stimulation described above. Both interventions will be administered simultaneously over an 8-week period, in accordance with the respective protocols.
  Interventions: Other: VR+OKS

INTERVENTIONS:
Other: Optokinetic Virtual Reality Stimulation — The optokinetic stimulation protocol is defined as follows:
  * Optokinetic stimulation sessions are planned with a balloon rotation speed of 20°/s (degrees per second) during the first four weeks. In the fifth and sixth weeks, the speed will be increased to 25°/s, and in the seventh and eighth weeks, it will be raised to 30°/s.
  * The background screen will be set to rotate in the same direction as the balloons, with a rotation speed equal to 30-50% of the balloon rotation speed.
  * Session duration will start at 30 seconds and will increase to 150 seconds depending on patient tolerance as the sessions progress.
  * Participants will be instructed to focus on the red balloon in a moving visual scene.
  Optokinetic stimuli will be applied to participants in various postures: sitting, upright posture (feet together), semi-tandem stance, or tandem stance positions.
  Arms: Group 2 (OKS Group)
Other: Conventional rehabilitation program based on Cawthorne Cooksey exercises — The program will consist of Tracking, VOR, Neck, Static-Dynamic Balance Exercises and Walking training. These exercises depend on the patient's condition; It will be done in sitting, Romberg, semitandem, tandem and walking positions with eyes open and closed. Hard and soft grounds will be used.
  Arms: Group 1 (VR Group)
Other: VR+OKS — The optokinetic stimulation protocol is defined as follows:
  Optokinetic stimulation will be applied over 8 weeks with gradually increasing balloon rotation speeds: 20°/s (weeks 1-4), 25°/s (weeks 5-6), and 30°/s (weeks 7-8). The background will rotate in the same direction at 30-50% of the balloon speed. Sessions will start at 30 seconds and increase to 150 seconds based on tolerance. Participants will focus on a red balloon in a rotating visual scene, and the stimulation will be performed in various postures including sitting, feet together, semi-tandem, and tandem stance.
  The program will consist of Tracking, VOR, Neck, Static-Dynamic Balance Exercises and Walking training. These exercises depend on the patient's condition; It will be done in sitting, Romberg, semitandem, tandem and walking positions with eyes open and closed. Hard and soft grounds will be used.
  Arms: Group 3 (VR+OKS Group)

SUMMARY:
The study will be conducted on patients diagnosed with UVH who apply to Prof. Dr. Mete İşeri Ear, Nose and Throat Diseases Polyclinic and Güneşli Erdem Hospital Ear, Nose and Throat and Vestibular Rehabilitation Unit. Participants will be divided into 3 groups by simple randomization (closed envelope) method. To the vestibular rehabilitation group; A conventional rehabilitation program based on structured Cawthorne Cooksey exercises will be applied for 45 minutes once a week with the support of a physiotherapist for 8 weeks. To the optokinetic stimulation group; optokinetic stimulation will be given with virtual reality glasses, and to the combined group; Participants in the vestibular exercise group will receive additional optokinetic stimulation. The application will be done once a week for 8 weeks. Inclusion criteria for the study are; diagnosed with unilateral vestibular hypofunction with VNG test, between the ages of 18-65, class A+ in the System Usability Scale (SUS) and the percentage range being between 96-100%; Exclusion criteria for the study are; Bilateral vestibular hypofunction, visual impairment, neurological disorder and inability to communicate.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral vestibular hypofunction with VNG test,
* Being between the ages of 18-65,
* Being in the A+ class on the System Usability Scale (SCS) and having a value between 96-100 percentile

Exclusion Criteria:

* Having bilateral vestibular hypofunction
* Having a visual impairment,
* Having a neurological disorder
* Inability to communicate

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2025-09-07 (Estimated); Primary Completion 2025-10-07 (Estimated); Study Completion 2026-10-07 (Estimated)

PRIMARY OUTCOMES:
Headache Impact Scale (HIT-6): | 8 Weeks
  Bayliss et al. It is a short questionnaire designed to assess migraine pain from the patient's perspective and track lost time. Each item is answered using a 5-point Likert scale (6=never, 8=rarely, 10=sometimes, 11=very often, 13=always). The final score is determined from the sum of 6 items with a range from 36 to 78. Higher scores indicate greater impact.
Motion Sickness Severity Scale (MSSS) | 8 Weeks
  It is a 7-point scale rated from 0 to 6, where participants select the item that best describes their current condition: none (0), stomach awareness or discomfort (1), mild nausea (2), moderate nausea (3), severe nausea (4). ), gagging (5) or vomiting (6).
Simulator Sickness Survey (SHA) | 8 Weeks
  It has been widely used to evaluate various forms of disease triggered by virtual environments. 16 symptoms such as eye fatigue, nausea, sweating and headache are evaluated in 4 different severity levels (0: none, 1: mild, 2: moderate and 3: severe). Symptoms are grouped into 3 non-mutually exclusive categories representing nausea, oculomotor disturbance, and disorientation. Higher scores in each category indicate stronger perceptions of underlying disease symptoms. A total score above 20 is considered "poor-failing".

SECONDARY OUTCOMES:
Fatigue Severity Scale (FSS) | 8 Weeks
  It is a 7-point scale rated from 0 to 6, where participants select the item that best describes their current condition: none (0), stomach awareness or discomfort (1), mild nausea (2), moderate nausea (3), severe nausea (4), retching (5), or vomiting (6).
Dizziness Handicap Inventory (DHI) | 8 Weeks
  It is used to determine the physical, sensory and functional effects of vestibular system pathologies. Questions 1, 4, 8, 11, 13, 17 and 25: Physical disability; Questions 2, 9, 10, 15, 18, 20, 21, 22 and 23 examine emotional disability; Questions 3, 5, 6, 7, 12, 14, 16, 19 and 24: Refers to functional disability. For each question, the answers consist of yes (4 points), no (0 points) and sometimes (2). In scoring the subunits of the inventory, 28 points were accepted as the cut-off value to determine physical disability and 36 points to determine functional and sensory disability. High scores indicate that the patient's complaint of dizziness is severe.

OTHER OUTCOMES:
Sociodemographic data form | 8 Weeks
  In this form; The patient's age, gender, profession, whether he/she smokes and drinks alcohol, additional diseases, previous surgeries, medications used, history of the disease, onset of the disease, etc. will be questioned.

CONTACTS AND LOCATIONS:
Locations (1):
- Kocaeli Health and Technology University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No